CLINICAL TRIAL: NCT01794104
Title: A Phase I Trial of Weekly Indenoisoquinoline LMP400 in Adults With Relapsed Solid Tumors and Lymphomas
Brief Title: Indenoisoquinoline LMP400 for Advanced Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130080; 13-C-0080
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2017-10-27

CONDITIONS: Neoplasm; Lymphoma
Keywords: Topoisomerase Inhibitor; Advanced Malignancies; Pharmacodynamics; DNA Damage; Pharmacokinetics
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — NSC 724998

ARMS (1):
- 1 (Experimental): Open-label Phase I trial evaluating weekly administration of LMP400, on days 1, 8, and 15, in 28-day cycles.
  Interventions: Drug: LMP400

INTERVENTIONS:
Drug: LMP400 — Top1 inhibitors such as LMP400 are potent anticancer agents because stabilizing cleavage complex formation induces replication-and transcription-mediated DNA damage and delays DNA repair, leading to apoptosis. Preclinical and clinical data indicate that baseline tumor levels of Top1 correlate strongly with ability to respond to Top1 inhibitor therapy.

SUMMARY:
Background:

- Indenoisoquinoline LMP400 is an experimental cancer treatment drug. It damages DNA in tumor cells. Tumor cells with damaged DNA may die, resulting in cell death. Researchers want to see if this drug is a safe and effective treatment for solid tumors and lymphomas that have not responded to earlier treatment.

Objectives:

- To see if Indenoisoquinoline LMP400 is a safe and effective treatment for advanced solid tumors or lymphomas.

Eligibility:

- Individuals at least 18 years of age who have solid tumors or lymphomas that have not responded to treatment.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Tumor samples may also be collected. The size and location of the tumors will be determined with imaging studies.
* Indenoisoquinoline LMP400 is given in a 28-day cycle. Participants will receive the drug by intravenous infusion on days 1, 8, and 15 of each cycle, followed by a break of 13 days without the drug.
* Treatment will be monitored with frequent blood tests and imaging studies. Tumor samples will be optional.
* Participants will continue their cycles of treatment as long as the cancer does not grow and there are no severe side effects.

DETAILED DESCRIPTION:
Background:

* Indenoisoquinolines are non-camptothecin topoisomerase (Top1) inhibitors that form stable DNA-Top1 cleavage-complexes, have a preference for unique DNA cleavage sites, and are active against camptothecin-resistant cell lines. Unlike camptothecins, indenoisoquinolines are chemically stable and active in cells that over-express ATP-binding cassette (ABC) transporters ABCG2 and multidrug resistance (MDR-1). Top1 inhibitors are potent anticancer agents because stabilizing cleavage complex formation induces replication-and transcription-mediated DNA damage and delays DNA repair, leading to apoptosis. Preclinical and clinical data indicate that baseline tumor levels of Top1 correlate strongly with ability to respond to Top1 inhibitor therapy.
* A first-in-human Phase I study conducted at the NCI of the indenoisoquinoline LMP400 (NSC 743400) on a QD x 5 q28 schedule in patients with refractory solid tumors and lymphomas (10-C-0056) established that this agent is well tolerated. LMP400 shows linear pharmacokinetics with evidence of drug accumulation following 5 days of dosing. We hypothesize that weekly dosing (days 1, 8, 15 q28-day cycle) will increase LMP400 peak levels and exposures, improving clinical activity and safety.

Primary Objectives:

* To establish the safety and tolerability of weekly (days 1, 8, 15 q28-day cycle) LMP400 in patients with refractory solid tumors and lymphomas.
* To establish the maximum tolerated dose (MTD) of weekly LMP400 in patients with refractory solid tumors and lymphomas.
* To evaluate the pharmacokinetic profile of weekly LMP400.

Secondary Objectives:

* Evaluate the level of Top1 in tumor biopsies pre- and post- administration of LMP400.
* Evaluate the effect of LMP400 on markers of DNA damage and apoptosis, such as >=H2AX and caspase 3, in tumor biopsies pre- and post- LMP400 administration.

Eligibility:

-Patients with histologically confirmed metastatic solid tumors and lymphomas; adequate organ function.

Study Design:

* This is an open-label Phase I trial evaluating weekly administration of LMP400, on days 1, 8, and 15, in 28-day cycles.
* Starting dose is based on the MTD determined from the QD x 5, q28 day schedule currently being evaluated. The study will follow a 3 plus 3 design.
* Once the MTD is established, 10 additional patients will be enrolled at the MTD to further define the pharmacokinetics and evaluate effect of study drug on DNA damage and apoptosis.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically-documented (confirmed at the Laboratory of Pathology, NCI), solid tumor malignancy, or Hodgkin's disease/non-Hodgkin lymphoma, that is metastatic or unresectable and for which standard curative measures do not exist or are associated with minimal patient survival benefit.
* The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Life expectancy >3 months.
* Patients must have normal or adequate organ and marrow function as defined below:

  * Leukocytes greater than or equal to 3,000/mcL
  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin less than or equal to 2.0 x institutional upper limit of normal (we will allow patients with Gilbert s syndrome with total bilirubin up to 2.5 mg/dL)
  * AST (SGOT)/ALT (SGPT) less than or equal to 3 x institutional upper limit of normal

    ---patients with metastatic disease in the liver less than or equal to 5 x ULN
  * Creatinine <1.5 x upper limit of normal
  * OR
  * Creatinine clearance

    * greater than or equal to 60 mL/minute for patients with creatinine levels
    * greater than or equal to 1.5 x institutional upper limit of normal
* Age greater than or equal to 18
* The effects of indenoisoquinolines on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months after completion of indenoisoquinolines administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of indenoisoquinolines administration
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients must have recovered to at least eligibility levels due to adverse events (AEs) and/or toxicity of prior chemotherapy or biologic therapy. They must not have had major surgery, chemotherapy, radiotherapy, or biologic therapy within 3 weeks (6 weeks for nitrosoureas and mitomycin C, or 2 months for UCN-01). Patients must be greater than or equal to2 weeks since any investigational agent administered as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a subtherapeutic dose of drug is administered) at the PI s discretion, and should have recovered to eligibility levels from any toxicities. However, patients receiving bisphosphonates for any cancer or undergoing androgen deprivation therapy for prostate cancer are eligible for this therapy. Prior therapy with topoisomerase I inhibitors is allowed.
* Patients who are receiving any other investigational agents.
* Patients with known active brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with brain metastasis stable for at least 4 weeks following surgery and/or radiation are eligible.
* Uncontrolled incurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with LMP400. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

INCLUSION OF WOMEN AND MINORITIES:

- Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02-15; Primary Completion 2016-05-19 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
To establish the safety and tolerability of weekly (days 1, 8, 15 q28-day cycle) LMP400 in patients with refractory solid tumors and lymphomas | Cycle 1

SECONDARY OUTCOMES:
Evaluate the level of Top1 in tumor biopsies pre and post- administration of LMP400 | Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Champoux JJ. DNA topoisomerases: structure, function, and mechanism. Annu Rev Biochem. 2001;70:369-413. doi: 10.1146/annurev.biochem.70.1.369. PMID 11395412
- [Background] Wang JC. Cellular roles of DNA topoisomerases: a molecular perspective. Nat Rev Mol Cell Biol. 2002 Jun;3(6):430-40. doi: 10.1038/nrm831. PMID 12042765
- [Background] Pommier Y. Topoisomerase I inhibitors: camptothecins and beyond. Nat Rev Cancer. 2006 Oct;6(10):789-802. doi: 10.1038/nrc1977. PMID 16990856
- [Derived] Beumer JH, Kennard BC, Holleran JL, Moore N, Zlott J, Miller BM, Kummar S, Chen A, Doroshow J, Park W, Gobburu J, Dunn A. Evaluating the indotecan-neutropenia relationship in patients with solid tumors by population pharmacokinetic modeling and sigmoidal Emax regressions. Cancer Chemother Pharmacol. 2023 Mar;91(3):219-230. doi: 10.1007/s00280-023-04509-8. Epub 2023 Feb 23. PMID 36813886